CLINICAL TRIAL: NCT07270315
Title: Effects of Self-Compassion on Reducing Problematic Gaming and Its Underlying Mechanisms: A Randomized Controlled Trial
Brief Title: Self-Compassion and Problematic Gaming: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, li,xinyi, Co-Investigator, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNU-poslab-IGD-2025; 202304140074 (Other: Institutional Review Board of the Faculty of Psychology, Beijing Normal University); 202304140075 (Other: Institutional Review Board of the Faculty of Psychology, Beijing Normal University)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Problematic Gaming; Self-Compassion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention Group (Experimental): Participants in this group received a 14-day online course titled Positive Self, designed to enhance self-compassion. The course included 14 didactic videos (approximately 10 minutes each) on self-compassion concepts and applications, as well as 14 guided audio meditations (approximately 6 minutes each). The meditation practice involved in this intervention began with 3 days of breathing meditation, followed by 11 days of loving-kindness meditation. This intervention has been shown to effectively promote self-compassion in prior research.
  Interventions: Behavioral: Positive Self - 14-Day Online Self-Compassion Course
- Waitlist Control Group (No Intervention): Participants in this group received no intervention during the 14-day study period and were instructed to refrain from engaging in other meditation or mindfulness practices. They completed the same pretest, posttest, and one-month follow-up assessments as the intervention group. After the study concluded, participants in this group were offered access to the Positive Self online self-compassion course.

INTERVENTIONS:
Behavioral: Positive Self - 14-Day Online Self-Compassion Course — The Positive Self intervention is a 14-day online course designed to enhance self-compassion. The course includes 14 didactic videos (approximately 10 minutes each) on self-compassion concepts and applications, along with 14 guided audio meditations (approximately 6 minutes each). The meditation practice involves breathing meditation for the first 3 days, followed by 11 days of loving-kindness meditation. This intervention has been shown to effectively promote self-compassion in previous research.
  Arms: Self-Compassion Intervention Group

SUMMARY:
This study investigates the impact of self-compassion on reducing problematic gaming behaviors among young adults. Problematic gaming has been linked to anxiety, depression, and social dysfunction, and this study aims to assess how self-compassion can address these issues. The study explores the role of basic psychological needs and social anxiety as mediators in this process.

A randomized controlled trial was conducted with 308 online game players (M = 22.40, SD = 3.52), who were randomly assigned to either an intervention group (n = 194) or a waitlist group (n = 114). The intervention consisted of an online self-compassion program. Participants completed pretest, posttest, and follow-up questionnaires to assess the changes in self-compassion and problematic gaming behaviors. The results indicated that the intervention significantly increased self-compassion and reduced problematic gaming through the same mediating pathways of basic psychological needs and social anxiety.

These findings suggest that self-compassion training may be an effective intervention for reducing problematic gaming behaviors among young adults, with implications for mental health interventions in gaming communities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older.
* Any gender.
* Recruited through online platforms.
* No restriction on educational background.
* Participants who regularly engage in online gaming and are willing to reduce or modify their gaming behaviors.

Exclusion Criteria:

* Individuals under 18 years old or those lacking full civil capacity.
* Individuals with diagnosed psychiatric or psychological disorders.
* Individuals without problematic gaming behaviors or without a clear intention to change their gaming habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Change in problematic gaming behavior score after 14-day self-compassion intervention | Baseline, post-intervention (Day 14), and one-month follow-up
  Participants' problematic gaming behavior was measured with an eight-item questionnaire adapted from Yang and Zhou (2004), a scale with established reliability and validity in Chinese samples. To match the intervention context, the term "video games" in the original items was replaced with "Genshin Impact" while maintaining the original semantic meaning. Items were rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree; α = .82). Higher scores reflected more severe problematic gaming behavior.

SECONDARY OUTCOMES:
Change in self-compassion score after 14-day self-compassion intervention | Baseline, post-intervention (Day 14), and one-month follow-up
  Participants' self-compassion was measured using the 12-item Short Form of the Self-Compassion Scale (Raes et al., 2011). The validated Chinese version (Chen et al., 2011) was used in this study. Items were rated on a 5-point Likert scale (1 = almost never, 5 = almost always; α = .84). Six items were reverse-scored. Higher total scores reflected greater levels of self-compassion.
Change in basic psychological needs score after 14-day self-compassion intervention | Baseline, post-intervention (Day 14), and one-month follow-up
  Participants' satisfaction of basic psychological needs was assessed using a 21-item questionnaire (Gagné, 2003; Liu et al., 2013). Items were rated on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree; α = .88). Nine items were reverse-scored. Higher scores reflected greater fulfillment of basic psychological needs.
Change in social anxiety score after 14-day self-compassion intervention | Baseline, post-intervention (Day 14), and one-month follow-up
  Participants' social anxiety was assessed using the 17-item Social Phobia Inventory. Items were rated on a 5-point scale (0 = not at all, 4 = extremely; α = .82). Higher scores reflected greater severity of social anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding sharing individual participant data (IPD) has not yet been finalized. Data may be shared in de-identified form after publication, depending on ethical approval and institutional policies at that time.